CLINICAL TRIAL: NCT00316225
Title: A Phase 2 Study of ALIMTA in Solid Tumor Patients With Stable Third-Space Fluid
Brief Title: Study of Pemetrexed in Mesothelioma and Lung Cancer Patients With Fluid Around the Lungs or Abdomen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10426; H3E-MC-JMHX (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Results first posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-06

CONDITIONS: Non-small Cell Lung Cancer; Mesothelioma; Lung Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma; Lung Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed (Experimental): Pemetrexed 500 mg/m^2 intravenous (IV) every 21 days for 6 cycles
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 500 milligrams per meter squared (mg/m^2) IV every 21 days for 6 cycles
  Other Names: LY231514; Alimta

SUMMARY:
This study will test the effects of pemetrexed on mesothelioma and non-small cell lung cancer patients with fluid around their lungs or abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic (Stage III or IV at entry) non-small cell lung cancer (NSCLC) or mesothelioma
* Presence of third-space fluid (fluid around the lungs or abdomen).
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Prior anticancer treatment (except radiation) must be completed at least 3 weeks prior to study enrollment, and the patient must have recovered from the sharp toxic effects the anticancer treatment.
* Estimated life expectancy of at least 8 weeks.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that was not a marketed product.
* Active infection that, in the opinion of the investigator, would not allow the patient to tolerate therapy.
* Pregnancy.
* Breast-feeding.
* Significant weight loss (that is, greater than or equal to 10% of body weight) over the 6 weeks before study entry.
* Brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Copenhagen, Denmark
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid, Spain

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed: Pemetrexed 500 mg/m2 intravenous (IV) every 21 days for 6 cycles
Period: Overall Study
Arm/Group | Pemetrexed
Started | 31
Completed | 6
Not Completed | 25
Not completed — Adverse Event | 2
Not completed — Physician Decision | 3
Not completed — Progressive Disease | 15
Not completed — Withdrawal by Subject | 3
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
Age Continuous [Median (Full Range); unit: years] | 62.7 [35.7 to 77.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 30
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  Spain | 12
  Denmark | 6
  Germany | 13
Diagnosis [Number; unit: participants] — Diagnosis of Non-Small Cell Lung Cancer (NSCLC) and mesothelioma were determined by each individual investigator.
  participants
    Non-Small Cell Lung Cancer (NSCLC) | 23
    Mesothelioma | 8
Disease Stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body).
  participants
    Stage III (locally advanced disease) | 12
    Stage IV (metastatic disease) | 18
    Unknown | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 14
    1 - Ambulatory, Restricted Strenuous Activity | 17
Fluid Severity [Number; unit: participants] — Mild = (1) pleural effusion detectable on radiological imaging, but less than moderate; (2) ascites detectable only by radiological imaging. Moderate = (1) pleural effusion less than 1/3 of the way up the thorax on 1 side on imaging and obscuring the entire hemidiaphragm on that side; (2) ascites detectable on physical exam (that is, fluid wave is palpable). Severe = (1) pleural effusion more than 1/3 of the way up the thorax on imaging; (2) ascites visibly detectable.
  For Moderate Fluid Severity, there were 13 patients with pleural effusion and 1 patient with ascites.
  participants
    Mild | 15
    Moderate | 14
    Severe | 2
Primary Basis for Diagnosis [Number; unit: participants]
  Cytological | 6
  Histopathological | 25
Type of Third-Space Fluid [Number; unit: participants]
  Pleural Effusion | 30
  Ascites | 1
Body Surface Area [Median (Full Range); unit: meters squared (m^2)] | 1.8 [1.4 to 2.3]
Height [Median (Full Range); unit: centimeters (cm)] | 171.0 [147.0 to 189.0]
Weight [Median (Full Range); unit: kilograms (kg)] | 68.0 [47.9 to 100.0]

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Common Toxicity Criteria - National Cancer Institute Grade 3 and Grade 4 Toxicities
Description: Number of participants with laboratory and non-laboratory toxicities possibly related to study drug, which were graded using the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) for defining and grading specific adverse events. Grades range from 0 (none) to 5 (death). Grade 3 is severe and Grade 4 is life-threatening.
  NOS = Not otherwise specified.
Time Frame: baseline, up to 18 weeks
Population: Patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
participants
  Leukocytopenia | 1
  Neutropenia/Granulocytopenia | 1
  Platelets | 1
  Ascites (Non-Malignant) | 1
  Febrile Neutropenia | 1
  Pain Pulmonary/Upper Respiratory-Chest/Thorax NOS | 1
  Pleural Effusion (Non-Malignant) | 1

2. Secondary Outcome: Pemetrexed Population Pharmacokinetics (PK): Clearance
Description: Clearance (CL) can be defined as the volume of plasma which is completely cleared of drug (pemetrexed) per unit time. Total body clearance is calculated after intravenous administration of the drug (pemetrexed) and is measured by taking plasma samples at various timepoints and measuring the amount of pemetrexed in the plasma.
Time Frame: Cycle 1 and Cycle 2: before the end of infusion (approximately 9.5 minutes), 2 hours, 9-10 hours, 24-48 hours, 480-528 hours (20 to 22 days) after start of pemetrexed infusion
Population: Patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: milliliter per minute (mL/min)
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
milliliter per minute (mL/min) | 85.6 (21.4)

3. Secondary Outcome: Pemetrexed Population Pharmacokinetics: Volume of Distribution
Description: Volume of distribution is the theoretical size of the compartment necessary to account for total drug amount in the body if it were present throughout the body in the same concentration found in plasma. Volume of distribution is defined as distribution of pemetrexed in the body and is determined by volume of distribution = dose/drug concentration. By knowing dose and measuring concentration of pemetrexed in plasma, volume was calculated. Central volume (V1) was determined by dose/peak serum level of pemetrexed. Peripheral volume (V2) is sum of all tissue spaces outside the central compartment.
Time Frame: as for outcome 2
Population: Patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
Liters (L)
  Central Volume of Distribution | 6.61 (1.32)
  Peripheral Volume of Distribution (V2) | 8.91 (1.68)
  Peripheral Volume of Distribution (V3) | 1.26 (0)

4. Other Pre Specified Outcome: Overall Tumor Response
Description: Overall tumor response was determined using Response Evaluation Criteria In Solid Tumors (RECIST), which defines when cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments.
  CR (complete response) = disappearance of all target lesions. PR (partial response) = 30% decrease in the sum of the longest diameter of target lesions.
  PD (progressive disease) = 20% increase in the sum of the longest diameter of target lesions.
  SD (stable disease) = small changes that do not meet above criteria.
Time Frame: baseline, up to 18 weeks
Population: Patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 8
  Progressive Disease | 12
  Unknown | 9

5. Secondary Outcome: Discontinuations Due to Adverse Events
Description: Adverse events were coded using the Medical Dictionary for Regulatory Activities, Version 11.0.
Time Frame: baseline, up to 18 weeks
Population: Patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
participants
  Atrial fibrillation | 1
  Febrile neutropenia (possibly related) | 1
  Pneumonia (resulted in death) | 1
  Respiratory failure (resulted in death) | 1

6. Primary Outcome: Overview of Adverse Events
Description: Any untoward medical occurrence in a patient who received study drug was considered an adverse event (AE), without regard to possibility of causal relationship. Treatment-emergent adverse events (TEAE): those which occurred or worsened after baseline. An adverse event resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a serious adverse event (SAE): death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: baseline, up to 18 weeks
Population: Patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 31
participants
  TEAE - All, regardless of causality | 28
  TEAE - Possibly related to study drug | 23
  SAE - All, regardless of causality | 12
  SAE - Possibly related to study drug | 1
  Discontinuations Due to SAEs (including death) | 4
  Discontinuations - Possibly related to study drug | 1
  Discontinuations Due to Nonserious AEs | 0
  Deaths - On Study | 2
  Deaths - Possibly related to study drug | 0
  Deaths - Within 30 days of Study Discontinuation | 0

ADVERSE EVENTS:
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 12/31
Other Adverse Events (participants affected / at risk) | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (3)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pericardial excision (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed (N=31)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (11)
Vomiting (Gastrointestinal disorders) | 3 (4)
Asthenia (General disorders) | 8 (11)
Chest pain (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (13)
Influenza like illness (General disorders) | 2 (2)
Mucosal inflammation (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 5 (5)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 3 (9)
Respiratory tract infection (Infections and infestations) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days